CLINICAL TRIAL: NCT03134040
Title: Using Behavioral Economics to Promote Exercise Among Overweight Inactive Adults
Brief Title: Small Monetary Incentives to Promote Exercise (Exercise4Good; EX4G)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CA188473-02
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Physical Activity
Keywords: Incentives; Motivation
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Incentives (Rebate) (Experimental): On a weekly basis, participants receive a small monetary incentive to exercise each time they attend the YMCA.
  Interventions: Behavioral: Incentives (Rebate)
- Incentives (Donation) (Experimental): On a weekly basis, a small monetary incentive to exercise is provided in the form of a donation to a charity of the participant's choice for attendance at the YMCA.
  Interventions: Behavioral: Incentives (Donation)
- Control (Active Comparator): Participants receive feedback on their exercise attendance on a weekly basis.
  Interventions: Behavioral: Feedback

INTERVENTIONS:
Behavioral: Incentives (Rebate)
  Arms: Incentives (Rebate)
Behavioral: Incentives (Donation)
  Arms: Incentives (Donation)
Behavioral: Feedback
  Arms: Control

SUMMARY:
This study is for physically inactive adults with an active membership at a Greater Providence Young Men's Christian Association (YMCA).

Participants will receive weekly feedback on their attendance at the YMCA, and will be enrolled in the study for 1 year.

Participants will be assigned to one of three conditions, to either receive weekly: (i) monetary incentives, (ii) donations to a charity of their choice, or (iii) feedback only.

In order to continue to receive incentives, participants must maintain an active membership at the YMCA.

DETAILED DESCRIPTION:
The investigators propose to conduct a pilot study to test feasibility and proof-of-concept for two incentive programs to promote exercise among low-active overweight and obese adults. To address weaknesses in the literature, the programs will be (a) conducted in a community setting by the Greater Providence YMCAs and (b) financially sustainable, such that they do not require removal of the incentives after a specified period of time. In both incentive programs, participants will pay the standard monthly YMCA membership fee. In the Rebate incentive program, participants will have the opportunity to earn a small monetary incentive to exercise for each day that they attend the YMCA (verified by objective swipe-card data), with a maximum of 5 exercise sessions being incentivized per week. In the Donation incentive program, participants will have the opportunity to earn a small monetary incentive to exercise in the form of donations (using the same incentive schedule) to a registered local charity of the participant's choice. Thus, the proposed study will compare three experimental conditions: (a) Rebate incentives (n=25); (b) Donation incentives (n=25); and (c) Control (i.e., no incentives) (n=25). The Primary Aims are to test (1) feasibility of the two incentive programs, (2) feasibility of the research methods to evaluate the preliminary efficacy of the two incentive programs, and (3) proof-of-concept for the two incentive programs (relative to control), through comparison of average number of sessions/week with incentives over one year. Secondary outcomes will be self-reported minutes per week of exercise over one year. The proposed research will provide a preliminary investigation into two community-based, financially sustainable incentive programs to promote exercise for adults who are at increased risk for cancer. Positive findings from such a trial would provide a fast-track for a community-based ready-to-implement exercise promotion intervention. Additionally, such findings would have significant implications for the use of financially sustainable incentive programs for exercise through other community organizations (e.g., privately-owned health clubs), healthcare organizations, or employers (e.g., employer fitness facilities), as well as providing a model for incentive programs for other health-related behaviors (e.g., smoking cessation, weight loss).

ELIGIBILITY:
Inclusion Criteria:

* Inactive adults with an active YMCA membership
* Currently physically able to exercise

Exclusion Criteria:

* Do not plan to reside in the geographical region for the next 12 months
* Family member currently participating in the study
* Currently engaging in >150 mins of moderate/vigorous physical activity per week
* Attended the YMCA more than 4 times per month in the last 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Exercise attendance | 1 year
  How frequently the participant attended the YMCA during the study

CONTACTS AND LOCATIONS:
Overall Officials: David M Williams, PhD, Principal Investigator — Brown University; Omar Galarraga, PhD, Principal Investigator — Brown University
Locations (1):
- Public Health Building @ 121 South Main St, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with interested parties after all of the initial study analyses and outcomes have been published.
Time Frame: Data will be available 1 year after study completion.
Access Criteria: All data access requests will be reviewed by a panel prior to acceptance.

REFERENCES:
- [Derived] Galarraga O, Bohlen LC, Dunsiger SI, Lee HH, Emerson JA, Boyle HK, Strohacker K, Williams DM. Small sustainable monetary donation-based incentives to promote physical activity: A randomized controlled trial. Health Psychol. 2020 Apr;39(4):265-268. doi: 10.1037/hea0000818. Epub 2019 Nov 21. PMID 31750676